CLINICAL TRIAL: NCT07306026
Title: Evaluation of Toothbrush Bristles in Reduction of Plaque, Inflammation, Bleeding, and Abrasion: A Comparative Study of Tapered vs. End-Rounded Bristles
Brief Title: Evaluation of Toothbrush Bristles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Marcelle Nascimento, Assistant Dean for Clinical Research, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009358
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Gingivitis and Periodontal Diseases
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product A (Other): Product A: Double Tapered J-hook bristles (GUM® Technique® Deep Clean Toothbrush, 525 TPA1)
  Interventions: Other: Toothbrush with tapered bristles
- Product B (Other): End rounded bristles: (GUM® Technique® Deep Clean Toothbrush, 525 TPA1)
  Interventions: Other: Toothbrush with end-rounded bristles

INTERVENTIONS:
Other: Toothbrush with tapered bristles — Toothbrush with tapered bristles
  Arms: Product A
Other: Toothbrush with end-rounded bristles — Toothbrush with end-rounded bristles
  Arms: Product B

SUMMARY:
The goal of this randomized clinical trial is to investigate two different types of toothbrush bristles.

The main questions it aims to answer are the effects of two different bristle types on:

* how much plaque is on the teeth
* how deep the space is between gums and teeth
* how much gum and bone are attached to the teeth
* whether the gums bleed when checked
* if the gums get scratched or irritated

Researchers will compare toothbrushes with tapered bristles to those with regular round bristles.

Participants will be randomly assigned toothbrush A or B to use at home during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have read, understood and signed an informed consent prior to being entered into the study.
* Must be 18 to 70 years of age, male or female.
* Have at least 20 natural or restored teeth, not including implants.
* Must have average Plaque Index of greater than 2 at screening.
* Must have more than 20% of pockets with bleeding on probing at screening.
* Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures any time during the study.
* Agree to refrain from regular oral hygiene regimen for 24 hours and eating for 4 hours before the appointment in the study.
* Agree to abstain from the use of any dental products other than those provided in the study.
* Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

* Physical limitations or restrictions that might preclude normal tooth brushing.
* Evidence of gross oral pathology
* Periodontal probing pocket depths (PPD) ≥ 5mm.
* Evidence of major soft tissue lesions or trauma at the baseline visit as determined by the examiner.
* Chronic disease with concomitant oral manifestations
* Subjects who are currently undergoing, or require, extensive dental work, orthodontic treatment or periodontal surgery, or orthodontic treatment in the preceding 3 months
* Currently using bleaching trays
* Eating disorders
* Recent history of substance abuse
* Smoking >10 cigarettes/day
* Participation in other clinical studies within 14 days of screening
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Rustogi Modified Navy Plaque Index | Baseline, Week 2 and Week 4
  Measured before and after on-site brushing to compare the frequency of plaque presence before and after brushing, as well as cumulative effects of brushing over 2 and 4 weeks.

SECONDARY OUTCOMES:
Gingival Abrasion Score | Baseline, Week 2, and Week 4
  Measured before and after on-site brushing and categorized based on abrasion size (small, medium, large) to assess the one-time brushing effects as well as the cumulative effects of brushing over 2 and 4 weeks.

OTHER OUTCOMES:
Bleeding on Probing | Baseline, Week 2, Week 4
  Measured before and after on-site brushing to assess the one-time brushing effects as well as the cumulative effects of brushing over 2 and 4 weeks.
Periodontal Probing Depth and Clinical Attachment Loss | Baseline, Week 2 and Week 4
  PPD and CAL will be determined at six sites per tooth (mesio-facial, mid facial, disto-facial, disto-lingual, mid lingual, and mesio-lingual) to assess changes over 4 week study period.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Nascimento, DDS, MS, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- SUNY Buffalo School of Dental Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT07306026/Prot_SAP_000.pdf